CLINICAL TRIAL: NCT06951997
Title: Clinical Study on the Efficacy and Safety of Iparomlimab and Tuvonralimab Injection Combined With Chidamide, Albumin-bound Paclitaxel and Gemcitabine as First-line Treatment for Metastatic Pancreatic Cancer
Brief Title: QL1706 Plus Chidamide, AG as First-line Treatment for Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-PC-QIBA-3002
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706, Chidamide, Albumin-bound Paclitaxel and Gemcitabine (Experimental): QL1706 5mg/kg，Q3W; Gemcitabine 1000mg/m2 Q3W；Nab-paclitaxel 125mg/m2 Q3W; Chidamide, 20mg biw q3w;
  Interventions: Drug: QL1706; Drug: Chidamide; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: QL1706 — 5mg/kg, q3w
Drug: Chidamide — 20mg, biw, q3w
Drug: Gemcitabine — 1000mg/m2 Q3W
Drug: Nab-paclitaxel — 125mg/m2 Q3W

SUMMARY:
This is a single-center, open-label, exploratory study aims to assess the efficacy and safety of QL1706 plus nab-paclitaxel and gemcitabine as first-line treatment for patients with metastatic pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign the informed consent form for this study
* Age ≥18 years and ≤ 75 years, ale or Female
* Histologically or cytologically confirmed diagnosis of pancreatic cancer (originating from the pancreatic ductal epithelium), with clinical records showing metastatic pancreatic cancer (stage IV according to the AJCC 8th edition TNM staging of pancreatic cancer)
* No prior anti-tumor treatment (radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.) received
* At least one measurable lesion on imaging according to RECIST 1.1
* ECOG score 0-1
* Expected survival time ≥3 months
* Adequate organ function, subjects must meet the following laboratory criteria:Platelet count ≥90x10^9/L,White blood cell count ≥ 3.5 × 10⁹/L,Absolute neutrophil count (ANC) ≥1.5x10^9/L,Hemoglobin > 90g/L,Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN,Total bilirubin ≤ 1.5 ULN,Urea/Urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5 × ULN (and creatinine clearance rate (CCr) ≥ 50 mL/min),Left ventricular ejection fraction (LVEF) ≥ 50%,QTcF interval (Fridericia correction) < 470 ms
* Fertile women/non-sterilized men must use effective contraception

Exclusion Criteria:

* Inability to comply with the study protocol or procedures
* patients with pancreatic cancer originating from non-pancreatic ductal epithelium, including pancreatic neuroendocrine carcinoma, pancreatic follicular cell carcinoma, pancreatoblastoma, and solid-pseudopapillary tumors
* Known presence of germline BRCA1/2 mutations
* patients with known central nervous system metastases
* Hypersensitivity or allergic predisposition to the study drug or its excipients
* Concurrent use of any other investigational drug or participation in another clinical trial involving investigational therapy within 4 weeks
* Major surgery, severe traumatic injury, fractures, or ulcers within 6 weeks before study
* History of gastrointestinal perforation or fistula within 6 months before the first dose. Subjects may be enrolled if the perforation/fistula has been surgically repaired and the investigator confirms resolution
* Clinically significant gastrointestinal disorders, including obstruction (including partial), dysphagia, malabsorption syndrome, or uncontrolled nausea, vomiting, diarrhea, or other conditions severely affecting nutrient absorption
* Clinically significant bleeding or clear bleeding tendency within 1 month before the first dose, e.g.,gastrointestinal bleeding, hemorrhagic gastric ulcer
* Any of the following concurrent conditions:(1) Uncontrolled hypertension, coronary artery disease, arrhythmia, or heart failure(2) Severe uncontrolled concurrent infection causing disability(3) Proteinuria ≥ 2+ (≥1.0 g/24 h)(4) Bleeding tendency or history within 2 months before enrollment, regardless of severity(5) Arterial/venous thromboembolic events within 12 months before treatment (e.g., cerebrovascular accident, transient ischemic attack)(6) Acute myocardial infarction, acute coronary syndrome, or CABG within 6 months before treatment(7) Unhealed fractures or chronic wounds(8) Coagulopathy, bleeding tendency, or ongoing anticoagulation therapy
* History of other malignancies within 5 years before enrollment, except for adequately treated basal/squamous cell skin cancer or cervical carcinoma in situ
* Any cardiovascular or cerebrovascular disease or risk factors
* Active autoimmune disease or history of autoimmune disease within 4 weeks before enrollment
* Prior allogeneic bone marrow or solid organ transplantation
* Unresolved toxicities (> CTCAE v5.0 Grade 1) from prior anticancer therapy, except alopecia, lymphopenia, and oxaliplatin-induced neurotoxicity (≤ Grade 2)
* Prior treatment with immune checkpoint inhibitors (e.g., anti-PD-1/PD-L1/CTLA-4 antibodies), immune checkpoint agonists (e.g., anti-ICOS/CD40/CD137/GITR/OX40 antibodies), or immune cell therapy (e.g., CAR-T)
* Systemic treatment with corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressants within 14 days before the first dose
* Known interstitial lung disease (ILD) or non-infectious pneumonitis (either symptomatic or requiring systemic steroids)
* Any other clinically significant condition, metabolic disorder, physical/lab abnormality, epilepsy requiring treatment etal
* Pregnant or breastfeeding women
* Any other condition deemed unsuitable for study participation by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  overall response rate

SECONDARY OUTCOMES:
OS | 2 year
  OS is defined as the time from date of treatment start to the date of death from any cause or to the date of last follow-up if patients are alive. If a patient is alive by the time of final analysis, the patient will be censored at the last follow-up date.
AEs | 2 year
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0
Progression-free Survival (PFS) | 2 year
  PFS was assessed by investigators per RECIST 1.1
Disease Control Rate (DCR) | 2 year
  DCR was assessed by investigators per RECIST 1.1
Duration of Response (DOR) | 2 year
  DOR was assessed by investigators per RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China